CLINICAL TRIAL: NCT06471946
Title: Venetoclax Plus Azacytidine Conditioning Regimen Allo-HSCT for Elderly Patients With Higher-risk Myelodysplastic Syndromes
Brief Title: VA Conditioning Regimen Allo-HSCT for Elderly Higher-risk MDS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liren Qian, Vice Director, Navy General Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAHCT2024
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Higher-risk Myelodysplastic Syndromes
MeSH Terms: interventions — venetoclax

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venetoclax Plus Azacytidine Conditioning Regimen Allo-HSCT (Experimental): Patients were treated by Venetoclax Plus Azacytidine Conditioning Regimen Allo-HSCT
  Interventions: Drug: Venetoclax Plus Azacytidine Conditioning Regimen Allo-HSCT

INTERVENTIONS:
Drug: Venetoclax Plus Azacytidine Conditioning Regimen Allo-HSCT — Patients were treated by VA Conditioning Regimen Allo-HSCT:
  Venetoclax 100mg po qd d1, 200mg po qd d2, 400mg po qd d3-14; Azacytidine 75 mg/m2 subcutaneous injection qd d1-7, donor stem cells infused from d9
  Other Names: VA Conditioning Regimen Allo-HSCT

SUMMARY:
The goal of this phase 1/2 trial is to test the safety and efficacy of Venetoclax Plus Azacytidine Conditioning Regimen Allo-HSCT in treating patients with higher-risk MDS.

DETAILED DESCRIPTION:
The investigators will evaluate 2 year overall survival(OS) after transplantation in patients with higher-risk MDS. Progression free survival (PFS), incidence of acute GVHD, non-relapse mortality (NRM), graft-versus-host disease (GVHD)-free relapse-free survival(GRFS), and incidence of chronic GVHD at 1 and 2 years after transplantation will be counted.

ELIGIBILITY:
Inclusion Criteria:

* The patient should, in the investigator's opinion, be able to meet all clinical trial requirements.
* The patient is willing and able to adhere to the study visit schedule and other protocol requirements.
* The patient should be diagnosed with higher risk MDS according to the standard criteria of the World Health Organization (WHO).

Exclusion Criteria:

* Active or uncontrolled infections requiring systemic treatment within 14 days before enrollment.
* Any instability of systemic disease, including but not limited to severe cardiac, liver, kidney, or metabolic disease need therapy.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2029-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 3 year
  OS was defined as time from diagnosis to death from any cause or the last follow-up

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 3 year
  For patients in morphologic remission, documented relapse was considered progression.
Incidence of acute GVHD and chronic GVHD | 3 year
  Incidence rate of acute GVHD and chronic GVHD
Non-relapse mortality (NRM) | 3 year
  Non-relapse mortality (NRM) was defined as death from any cause not subsequent to relapse.
Graft-versus-host disease (GVHD)-free relapse-free survival(GRFS) | 3 year
  Graft-versus-host disease (GVHD)-free relapse-free survival(GRFS) was defined as petients without GVHD and relapse

CONTACTS AND LOCATIONS:
Overall Officials: Liren Qian, PhD, Principal Investigator — Navy General Hospital, Beijing
Locations (1):
- Navy General Hospital, Beijing, Beijing Municipality, China